CLINICAL TRIAL: NCT06863077
Title: The Evaluation of Knee Medial Collateral Ligament Recovery With Shear-Wave Elastography After Pie-Crusting Release Technique
Brief Title: Knee Medial Collateral Ligament Recovery After Pie-Crusting Release Technique
Status: Active, not recruiting | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Sabır, MD, Kastamonu University
Other Study IDs: 2024-KAEK-199
Record Dates: First submitted 2025-01-22; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Medial Collateral Ligament; Medial Mensical Tear; Shear Wave Elastography
Keywords: medial collateral ligament; pie-crusting; shear wave elastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pie-Crusting: MCL Pie-Crusting
  Interventions: Procedure: MCL Pie-Crusting

INTERVENTIONS:
Procedure: MCL Pie-Crusting — Percutaneous MCL Pie-Crusting

SUMMARY:
Medial meniscus tears requiring surgical interventions are mostly being done by arthroscopic procedures. During the arthroscopy, accessing the medial joint space is challenging. Because of this situation, pie-crusting of the medial collateral ligament (MCL) of the knee is described. This procedure is to release the MCL 1 cm distal to its origin with a needle-tip. This release provides enough space for both identifying the tear and also provides enough space to introduce necessary equipment in the joint space for repair. But there are some doubts about MCL release. Some authors suspected ongoing valgus instability after this procedure. Our aim is to identify the tension of MCL with USG shear wave elastography before the procedure, and 3 weeks, 6 weeks and 3 months postoperatively.

DETAILED DESCRIPTION:
Meniscal lesions are common orthopedic injuries. Posterior horn and medial meniscus root injuries are frequently seen as isolated cases or in association with ligament injuries ( 1 , 2 ). Arthroscopy is the preferred treatment method, and proper visualization of the medial compartment of the knee is crucial for correct diagnosis and treatment. Arthroscopic visualization of the posteromedial aspect of the knee may be difficult in patients with medial narrow knee joints and no ligament injuries ( 1 , 2 ); inadequate visualization may lead to treatment failure with persistent symptoms such as pain, crepitation, or locking of the joint. Femoral or tibial cartilage damage may occur during arthroscopy due to the narrowness of the medial compartment of the knee, due to the instruments used, which may lead to secondary osteoarthritis or to rupture of the medial collateral ligament (MCL) during valgus stress if excessive force is applied to open the medial joint space. During difficult manipulations, damage and breakage of arthroscopic instruments may occur. Therefore, in order to optimize imaging and intervention in medial knee joint pathologies, it is recommended to perform prophylactic controlled percutaneous needle-assisted loosening of the superficial medial collateral ligament during the operation (pie-crusting). However, there is a concern that the medial collateral ligament may not heal and laxity may develop. There are studies in the literature on patients who underwent medial collateral ligament loosening with the piecrusting method. In these studies, improvement has been shown in functional scores, physical examination (valgus stress), magnetic resonance imaging and knee valgus stress radiographs. However, the healing time and whether the medial collateral ligament has regained its former morphological characteristics have not been quantitatively demonstrated.

Share wave elastography uses sound waves to evaluate the mechanical properties of tissues such as stiffness and elasticity. They are used to detect different pathologies in tissues by using the differences in the mechanical properties mentioned above. Tissue stiffness is calculated using a physical property of tissue called Young's modulus or modulus of elasticity. Young's modulus is defined as the ratio of stress (force applied to the cross-sectional area of a given material) to strain (i.e., deformation; in this case, tissue deformation). The unit of Young's modulus is Pa (Pascal) or the SI unit is N/m2. The sonographic elastography value is usually in kPa (kilopascal) in most clinical settings. Patients who are scheduled for surgery with a diagnosis of medial meniscus tear will be evaluated ultrasonographically by 2 different radiologists in the preoperative period. Both knees will have medial collateral ligament share wave elastography performed and recorded. In patients who have undergone medial collateral ligament pie crusting for imaging of the knee medial compartment during the operation, share wave elastographic measurements will be performed by the same 2 radiologists again in the 3rd, 6th and 12th weeks after the operation. At the same time, the functional scores and examination findings of these patients in their outpatient clinic follow-ups will be noted. Preoperative and contralateral knee medial collateral ligament measurements of the patients will be used as the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Having a medial meniscus laceration detected in the magnetic resonance imaging taken due to the application for knee complaints and therefore having an indication for surgery
* Having consented to the surgical consent form explaining surgical and non-surgical options, accepting the surgical procedure
* Having consented to the research volunteer consent form presented to him/her verbally and in writing after giving his/her consent for surgery

Exclusion Criteria:

* Having had a previous fracture, meniscus tear, anterior or posterior cruciate ligament tear, medial or lateral collateral ligament tear in the same or opposite knee.
* Having had arthroscopic or open surgery around the knee due to or outside of the above reasons.
* Having had or not had surgery on the same lower extremity or the opposite lower extremity, having a fracture sequela or deformity.
* Having grade 1 or higher arthrosis according to the Kellgren-Lawrence arthrosis classification on direct radiographs taken before surgery.
* Patients who do not require medial collateral ligament release to access the medial joint space during surgery and therefore do not require pie-crusting medial collateral ligament release.
* Patients who wish to withdraw their consent given to the research volunteer consent form at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with medial meniscal injury
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MCL recovery | Preoperative and three months postoperative
  The shear wave elastography measured strain values of medial collateral ligament

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ali Sabır Sabır, M.D., Principal Investigator — Kastamonu University
Locations (1):
- Kastamonu Education and Research Hospital, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
During the writing process of the research, the age, operated side, preoperative value and postoperative follow-up values of shear wave elastographys are planned to be shared with the other researchers in the article.

REFERENCES:
- [Background] Herber AP, Brinkman JC, Tummala SV, Economopoulos KJ. Medial Collateral Ligament Pie-Crusting for Isolated Medial Meniscal Root Repair Is Associated With Improved Clinical Outcomes with Minimum 2-Year Follow-Up. Arthroscopy. 2024 Mar;40(3):869-875. doi: 10.1016/j.arthro.2023.07.029. Epub 2023 Jul 31. PMID 37532161
- [Background] Atoun E, Debbi R, Lubovsky O, Weiler A, Debbi E, Rath E. Arthroscopic trans-portal deep medial collateral ligament pie-crusting release. Arthrosc Tech. 2013 Jan 26;2(1):e41-3. doi: 10.1016/j.eats.2012.10.008. Print 2013 Feb. PMID 23802093